CLINICAL TRIAL: NCT02063893
Title: Study of Cancer Stem Cell Vcccinie That as a Specific Antigen in Metastatic Adenocarcinoma of the Breast
Brief Title: Safety Study of Cancer Stem Cell Vaccinie to Treat Breast Cancer
Acronym: CSC
Status: Completed | Type: Observational
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: CLB-001; 201401 (Other Grant/Funding Number: The research fund of Fuda cancer hospital in Guangzhou)
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will keep the CSC of every patient
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- non-vaccine
- giving low vaccine
- giving middle vaccine
- giving high vaccine

SUMMARY:
Most studies of cancer stem cells (CSC) involve the inoculation of cells from human tumors into immunosuppressed mice, preventing an assessment on the immunologic interactions and effects of CSCs. In this study, the investigators examined the vaccination effects produced by CSC-enriched populations from histologically distinctmurine tumors after their inoculation into different syngeneic immunocompetent hosts. Enriched CSCs were immunogenic and more effective as an antigen source than unselected tumor cells in inducing protective antitumor immunity.Immune sera from CSC-vaccinated hosts contained high levels of IgG which bound to CSCs, resulting in CSC lysis in the presence of complement.CTLs generated from peripheral blood mononuclear cells or splenocytes harvested from CSC-vaccinated hosts were capable of killing CSCs in vitro. Mechanistic investigations established that CSC-primed antibodies and T cells were capable of selective targeting CSCs and conferring antitumor immunity.

DETAILED DESCRIPTION:
To assess the feasibility of generating CSC-loaded DC vaccines for clinical use, the investigators will harvest peripheral blood and tumor specimen from patients with Breast Cancer. The investigators will purify T, B cells and generate DCs from the PBMCs of the Breast Cancer patient.On the other hand, investigators will isolate ALDHhigh and ALDHlow tumor cells from the tumor specimen of the Breast Cancer patient using a similar protocol as investigators reported .

Aim 1: To demonstrate, in vitro, the relative cellular anti-Breast Cancer CSC immunity induced by Breast Cancer CSC-DC primed cytotoxic T cells.

Aim 2: To determine, in vitro, specific binding and lysis of Breast Cancer CSCs by antibodies produced by purified B cells from PBMCs stimulated with Breast Cancer CSC-DC.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 30 years of age at the time the informed consent to screening has been obtained;
* The patient has one of the following histologically confirmed breast cancer subtypes:

Estrogen receptor and/or progesterone positive tumor; Human epidermal growth factor receptor 2 (HER2)-overexpressing breast cancer; HER2-negative breast cancer.

-- The patient shows normal organ function according to the following parameters(as measured within six weeks prior to treatment allocation):

* Hemoglobin: Within normal range according to institutional standards;
* Absolute leukocyte count: Within normal range according to institutional standards;
* Absolute lymphocyte count: Within normal range according to institutional standards;
* Platelet count: Within normal range according to institutional standards;
* Alanine aminotransferase: ≤ 2.5 x Upper Limit of Normal (ULN);
* Aspartate aminotransferase: ≤ 2.5 x ULN;
* Total bilirubin: ≤ 1.5 x ULN. In the case of known Gilbert's syndrome ≤ 2 x ULN;
* Serum creatinine: 1.5 x ULN;
* Calculated creatinine clearance: > 50 mL/min .

Exclusion Criteria:

* The patient has inflammatory breast cancer, which is defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion.
* Diagnosis established by incisional biopsy.
* Prior and concomitant neoadjuvant anti-breast-cancer treatments such as chemotherapy, immunotherapy / biological response modifiers, endocrine therapy, and radiotherapy, unless authorized specifically by the protocol.
* level 3 hypertension;
* severe coronary disease;
* myelosuppression;
* respiratory disease;
* brain metastasis;
* chronic infections

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who unresectable after Cryotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The primary study purpose to determine the safety of immunization with cancer stem cells vaccinie by the number of participants with adverse events | up to 3 months

SECONDARY OUTCOMES:
The secondary objectives are to evaluate vaccinie immune responses to the immunizations by the data of body measurements | 1 month

OTHER OUTCOMES:
The dose of CSC vaccine | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biological treatment center in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Ning N, Pan Q, Zheng F, Teitz-Tennenbaum S, Egenti M, Yet J, Li M, Ginestier C, Wicha MS, Moyer JS, Prince ME, Xu Y, Zhang XL, Huang S, Chang AE, Li Q. Cancer stem cell vaccination confers significant antitumor immunity. Cancer Res. 2012 Apr 1;72(7):1853-64. doi: 10.1158/0008-5472.CAN-11-1400. PMID 22473314
- See also: Related Info — http://www.fudahospital.com/